CLINICAL TRIAL: NCT00640471
Title: A Phase III Randomized Study of Brivanib Alaninate (BMS-582664) in Combination With Cetuximab (Erbitux®) Versus Placebo in Combination With Cetuximab (Erbitux®) in Patients With K-RAS Wild Type Tumors Previously Treated With Combination Chemotherapy for Metastatic Colorectal Carcinoma
Brief Title: Cetuximab With or Without Brivanib in Treating Patients With K-Ras Wild Type Tumours and Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CO20; CAN-NCIC-CO20 (Registry Identifier: NCI US - Physician Data Query); CDR0000590316 (Other: PDQ)
Record Dates: First submitted 2008-03-20; First posted 2008-03-21 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; brivanib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brivanib (Active Comparator)
  Interventions: Biological: cetuximab; Drug: brivanib alaninate
- Placebo (Active Comparator)
  Interventions: Biological: cetuximab

INTERVENTIONS:
Biological: cetuximab — cetuximab (Erbitux®) - Initial dose - Day 1 (Week 1): 400 mg/m2 IV over 120 minutes Maintenance Infusions (subsequent weeks): 250 mg/m2 IV over 60 minutes
Drug: brivanib alaninate — brivanib (BMS-582664) 800 mg po, QD
  Arms: Brivanib

SUMMARY:
RATIONALE: Brivanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether giving brivanib together with cetuximab is more effective than cetuximab alone in treating patients with metastatic colorectal cancer.

PURPOSE: This randomized phase III trial is studying cetuximab to see how well it works compared with cetuximab given together with brivanib in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the overall survival of patients with previously treated K-Ras wild type metastatic colorectal carcinoma treated with brivanib alaninate in combination with cetuximab versus placebo in combination with cetuximab.

Secondary

* To compare the progression-free survival of these patients.
* To compare the objective response rate and duration of response in these patients.
* To compare the quality of life of these patients.
* To compare the health utilities of these patients.
* To conduct a comparative economic evaluation of these patients.
* To evaluate the safety profile of this regimen in these patients.
* To explore an association between FGF-2, BRAF mutations, amphiregulin (AREG) and epiregulin (EREG) as determined from paraffin embedded tumor specimens and the potential for clinical benefit from the addition of brivanib alaninate or placebo to cetuximab in terms of overall survival, progression-free survival and objective response rate compared to cetuximab alone.
* To explore associations with mRNA and/or protein expression and/or variations in genes associated with epidermal growth factor (EGF), vascular endothelial growth factor (VEGF), angiogenesis, and other related pathways and the potential for clinical benefit from the addition of brivanib alaninate to cetuximab in terms of overall survival, progression-free survival, and objective response rate compared to cetuximab alone.
* To explore an association with changes of Collagen IV in the blood and the potential for clinical benefit from the addition of brivanib alaninate to cetuximab in terms of overall survival, progression-free survival and objective response rate compared to cetuximab alone.
* To establish a comprehensive tumor bank linked to a clinical database for the further study of molecular markers in colorectal cancer.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center and ECOG performance status (0-1 vs 2). Patients are randomized to 1 of 2 arms.

* Arm I: Patients receive oral brivanib alaninate once daily and cetuximab IV over 60-120 minutes once weekly.
* Arm II: Patients receive oral placebo once daily and cetuximab IV over 60-120 minutes once weekly.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Tumor tissue and blood samples are collected for correlative studies. Samples are analyzed for biomarker levels (Collagen IV, FGF-2, and epiregulin, amphiregulin, and BRAF mutation status) and correlation with response.

After completion of study treatment, patients are followed at 4 weeks and then every 8 weeks thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary colorectal cancer

  * Metastatic disease
* Tumor must be confirmed to be K-Ras wild type (i.e., No K-Ras mutation found) by means of mutation analysis performed on representative samples of diagnostic tumor tissue by a central reference laboratory (archival tumor samples are acceptable for K-Ras mutation analysis)
* Must have received a prior thymidylate synthase inhibitor (e.g., fluorouracil, capecitabine, raltitrexed, or tegafur-uracil) for adjuvant and/or metastatic disease

  * Thymidylate synthase inhibitor may have been given in combination with oxaliplatin or irinotecan hydrochloride
* Must meet one of the following criteria:

  * Received and failed* an irinotecan hydrochloride-containing regimen (i.e., single-agent or in combination) for treatment of metastatic disease
  * Relapsed within 6 months of completion of an irinotecan hydrochloride-containing adjuvant therapy
  * Has documented unsuitability** for an irinotecan hydrochloride-containing regimen NOTE: *Failure is defined as either progression of disease or intolerance to the irinotecan-containing regimen, where intolerance is defined as discontinuation due to any of the following: severe allergic reaction or delayed recovery from toxicity preventing retreatment NOTE: **Documented unsuitability for irinotecan includes known hypersensitivity to irinotecan, abnormal glucuronidation of bilirubin, Gilbert's syndrome, previous pelvic/abdominal irradiation, or elderly with comorbid conditions
* Must meet one of the following:

  * Received and failed* an oxaliplatin-containing regimen (i.e. single-agent or in combination) for treatment of metastatic disease
  * Relapsed within 6 months of completion of an oxaliplatin containing adjuvant therapy
  * Has documented unsuitability** for an oxaliplatin-containing regimen NOTE: *Failure is defined as either progression of disease or intolerance to the oxaliplatin-containing regimen, where intolerance is defined as discontinuation due to any of the following: severe allergic reaction, persistent severe neurotoxicity or delayed recovery from toxicity preventing retreatment

NOTE: **Documented unsuitability for oxaliplatin includes known hypersensitivity to oxaliplatin or other platinum compounds, pre-existing renal impairment, or Grade 2 or greater neurosensory neuropathy

* Measurable or evaluable disease
* Patient must consent to provision of, and investigator(s) must confirm access to and agree to submit at the request of the NCIC CTG Central Tumor Bank, a representative formalin fixed paraffin block of tumour tissue
* Patient must consent to provision of a sample of blood
* No symptomatic CNS metastases

  * Patients with signs or symptoms suggestive of brain metastasis are not eligible unless brain metastases are ruled out by CT or MRI scans

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2
* Absolute granulocyte count ≥ 1.5 x 10^9/L
* Platelet count ≥ 75 x 10^9/L
* Hemoglobin ≥ 80 g/L
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) (2.0 times ULN with documented liver metastases)
* ALT and AST ≤ 2.5 times ULN (5.0 times ULN with documented liver metastases)
* Serum creatinine ≤ 1.5 times ULN or creatinine clearance > 50 mL/min
* Magnesium > 0.5 mmol/L (1.2 mg/dL)
* LVEF > 45% by ECHO or MUGA scan
* No proteinuria ≥ 2+ on dipstick or ≥ 1 g on 24 hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to, during, and for 12 weeks after completion of study treatment
* Able (i.e., sufficiently fluent) and willing to complete the quality of life (EORTC QLQ-C30 and Skindex-16) and health utilities questionnaires (HUI3) in either English or French

Exclusion criteria:

* A history of other malignancies, except: adequately treated nonmelanoma skin cancer, curatively treated in situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years
* Any active disease condition which would render the protocol treatment dangerous or impair the ability of the patient to receive protocol therapy
* Any condition (e.g., psychological, geographical, etc.) that does not permit compliance with the protocol
* Uncontrolled or significant cardiovascular disease including any of the following:

  * Myocardial infarction within 12 months
  * Uncontrolled angina within 6 months
  * Clinically significant congestive heart failure
  * Stroke, transient ischemic attack, or other ischemic event within 12 months
  * Severe cardiac valve dysfunction
* Uncontrolled hypertension (consistent elevation of systolic BP > 150 and diastolic BP > 100 mmHg)
* History of a thromboembolic event in the last 6 months despite being treated with anticoagulation

  * Patients are eligible if they have experienced a thromboembolic event greater than 6 months previously and have initiated and are stable on anticoagulation or if they have previously initiated and are stable on anticoagulation for prevention of thromboembolic events
* Severe restrictive lung disease or radiological pulmonary findings of "interstitial lung disease" on the baseline chest x-ray which, in the opinion of the investigator, represents significant pathology
* Serious non-healing wounds, ulcers, or bone fractures
* History of allergy to brivanib (alaninate or related drug class
* Unable to swallow tablets

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Adequately recovered from recent surgery, chemotherapy and/or radiation therapy
* At least 4 weeks must have elapsed from major surgery, prior chemotherapy, prior treatment with an investigational agent or prior radiation therapy
* No prior cetuximab or other therapy* with targets the EGFR pathway (e.g., erlotinib hydrochloride, gefitinib hydrochloride, panitumumab)
* May have received a single prior regimen which targets the VEGFR pathway (e.g., bevacizumab , vatalanib, AZD2171, sorafenib tosylate, sunitinib malate, or others)
* No prior murine monoclonal antibody therapy (e.g., edrecolomab)
* No other concurrent chemotherapy
* No other concurrent therapies targeting the EGFR pathway (e.g., erlotinib, gefitinib, panitumumab, or others) or other therapies targeting the VEGFR pathway (e.g., bevacizumab , vatalanib, AZD2171, sorafenib tosylate, sunitinib malate, or others)
* Concurrent antihypertensive therapies allowed
* Concurrent aspirin allowed
* No other concurrent noncytotoxic experimental agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2008-05-12 (Actual); Primary Completion 2011-09-06 (Actual); Study Completion 2013-01-10 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years

SECONDARY OUTCOMES:
Progression-free survival | 3 years
Objective response rate | 3 years
Duration of response | 3 years
Quality of life (using EORTC QLQ-C30 and Skindex-16 Dermatology Survey) | 3 years
Health utilities (using HUI3 Health Utilities Index) | 3 years
Economic evaluation | 3 years
Safety profile | 3 years
Molecular markers | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lillian L. Siu, MD, FRCPC, Study Chair — Princess Margaret Hospital, Canada
Locations (37):
- Canada (37):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Abbotsford Centre, Abbotsford, British Columbia
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - The Vitalite Health Network - Dr. Leon Richard, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - The Royal Victoria Hospital, Barrie, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - PEI Cancer Treatment Centre,Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - L'Hotel-Dieu de Levis, Lévis, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quality of life (QoL) assessment in patients (pts) with K-RAS wild-type (WT) chemotherapy refractory metastatic colorectal cancer (mCRC) treated with cetuximab (CET) plus brivanib alaninate (BRIV) or placebo: Results of the NCIC Clinical Trials Group and AGITG CO.20 trial. J Clin Oncol 30, 2012 (suppl 4; abstr 542). Jolie Ringash, Heather-Jane Au, Lillian L. Siu, Jeremy D. Shapiro, Derek J. Jonker, John Raymond Zalcberg, Malcolm J. Moore, Andrew H. Strickland, Rami Kotb, Mark Jeffery, Thierry Alcindor, Siobhan Ng, Muhammad Salim, Sabe S. Sabesan, Jacob C. Easaw, Jennifer Anne Shannon, Fabyolla El-Tahche, Ian B. Walters, Dongsheng Tu, Christopher J. O'Callaghan.
- [Result] Phase III randomized trial of cetuximab (CET) plus either brivanib alaninate (BRIV) or placebo in patients (pts) with metastatic (MET) chemotherapy refractory K-RAS wild-type (WT) colorectal carcinoma (CRC): The NCIC Clinical Trials Group and AGITG CO.20 trial. J Clin Oncol 30, 2012 (suppl 4; abstr 386). Lillian L. Siu, Jeremy D. Shapiro, Derek J. Jonker, Christos Stelios Karapetis, John Raymond Zalcberg, John Simes, Felix Couture, Malcolm J. Moore, Timothy Jay Price, Jehan Siddiqui, Louise M. Nott, Danielle Charpentier, Winston S. Liauw, Michael B. Sawyer, Michael Jefford, Nadine M Magoski, Andrew Mark Haydon, Ian B. Walters, Dongsheng Tu, Christopher J. O'Callaghan.
- [Result] Final analysis of the phase III randomized trial of cetuximab (CET) plus either brivanib alaninate (BRIV) or placebo in patients (pts) with chemotherapy refractory, K-RAS wild-type (WT), metastatic colorectal carcinoma (mCRC): The NCIC Clinical Trials Group and AGITG CO.20 trial. J Clin Oncol 30, 2012 (suppl; abstr 3504). Lillian L. Siu, Jeremy David Shapiro, Derek J. Jonker, Christos Stelios Karapetis, John Raymond Zalcberg, John Simes, Felix Couture, Malcolm J. Moore, Timothy Jay Price, Jehan Siddiqui, Louise M. Nott, Danielle Charpentier, Winston S. Liauw, Michael B. Sawyer, Michael Jefford, Nadine M Magoski, Andrew Mark Haydon, Ian B. Walters, Dongsheng Tu, Christopher J. O'Callaghan.
- [Result] Analysis of plasma biomarkers potentially associated with antiangiogenic resistance in NCIC CTG/AGITG CO.20: A phase III randomized trial of cetuximab (CET) plus either brivanib alaninate (BRIV) or placebo in patients (pts) with chemotherapy refractory, k-RAS wild-type (WT), metastatic colorectal carcinoma (mCRC). J Clin Oncol 30, 2012 (suppl; abstr 3572). Jeremy David Shapiro, Lillian L. Siu, Christopher J O'Callaghan, John Raymond Zalcberg, Malcolm J. Moore, Timothy Jay Price, Catherine Doyle, John Simes, Brian Peter Findlay, Michelle F. Cronk, Asif Shaikh, Warren Lance Joubert, Benoit Samson, Antonino Bonaventura, Craig Underhill, David Wyld, Ian B. Walters, Penny Phillips, Dongsheng Tu, Derek J. Jonker.
- [Result] Siu LL, Shapiro JD, Jonker DJ, Karapetis CS, Zalcberg JR, Simes J, Couture F, Moore MJ, Price TJ, Siddiqui J, Nott LM, Charpentier D, Liauw W, Sawyer MB, Jefford M, Magoski NM, Haydon A, Walters I, Ringash J, Tu D, O'Callaghan CJ. Phase III randomized, placebo-controlled study of cetuximab plus brivanib alaninate versus cetuximab plus placebo in patients with metastatic, chemotherapy-refractory, wild-type K-RAS colorectal carcinoma: the NCIC Clinical Trials Group and AGITG CO.20 Trial. J Clin Oncol. 2013 Jul 1;31(19):2477-84. doi: 10.1200/JCO.2012.46.0543. Epub 2013 May 20. PMID 23690424
- [Derived] Nicholls DL, Xu MC, Zhan L, Sharma D, Hueniken K, Chiasson K, Wahba M, Brown MC, Grant B, Shapiro J, Karapetis CS, Simes J, Jonker D, Tu D, O'Callaghan C, Chen E, Liu G. Machine Learning Models of Early Longitudinal Toxicity Trajectories Predict Cetuximab Concentration and Metastatic Colorectal Cancer Survival in the Canadian Cancer Trials Group/AGITG CO.17/20 Trials. JCO Clin Cancer Inform. 2025 Apr;9:e2400114. doi: 10.1200/CCI.24.00114. Epub 2025 Apr 11. PMID 40215447
- [Derived] Hay AE, Pater JL, Corn E, Han L, Camacho X, O'Callaghan C, Chong N, Bell EN, Tu D, Earle CC. Pilot study of the ability to probabilistically link clinical trial patients to administrative data and determine long-term outcomes. Clin Trials. 2019 Feb;16(1):14-17. doi: 10.1177/1740774518815653. Epub 2018 Nov 22. PMID 30466310